CLINICAL TRIAL: NCT01879254
Title: Long-term Follow-up in Patients With Deep Brain Stimulation (DBS) for Severe Treatment Refractory Obsessive Compulsive Disorder (OCD).
Brief Title: Long-term Follow-up in Patients With Deep Brain Stimulation (DBS) for Obsessive Compulsive Disorder (OCD).
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s50928
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Obsessive Compulsive Disorder (OCD)
Keywords: obsessive compulsive disorder (OCD); deep brain stimulation (DBS); psychosurgery; long-term follow-up
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DBS for OCD
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation

SUMMARY:
For this human research, 17 treatment-refractory OCD patients who already received DBS implants for treatment refractory OCD between June 1998 and October 2007 will be included. New patients that complete the protocol on "refining the target for DBS in OCD" will be included in this follow-up study as well. They will be psychiatrically evaluated on regular bases: at least twice yearly in the years two to five after surgery, at least once a year for the years thereafter. The duration of this protocol is indefinite, but spans at least 10 years. The main aim of this study is to investigate the long-term effect of DBS in OCD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received DBS implantation for the treatment of OCD

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have received DBS for OCD will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2015-02-05 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium